CLINICAL TRIAL: NCT02742844
Title: An Interventional, Single Arm, Phase I/IIa Clinical Trial to Investigate the Efficacy and Safety of APZ2 on Wound Healing of Chronic Venous Ulcer (CVU)
Brief Title: Clinical Trial to Investigate Efficacy and Safety of the IMP in Patients With Non Healing Wounds Originating From Ulcers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID-19 pandemic and patient recruitment issues
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: Ticeba GmbH (Industry); FGK Clinical Research GmbH (Industry); Granzer Regulatory Consulting & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APZ2-II-01
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-02

CONDITIONS: Skin Ulcer Venous Stasis Chronic
Keywords: phase I/IIa; mesenchymal stem cells; ABCB5+; APZ2; chronic venous ulcer; varicose ulcer; skin ulcer; advanced therapy medicinal product; APZ2-II-01; autologous use; somatic cell therapy
MeSH Terms: conditions — Varicose Ulcer; Skin Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APZ2 application (Experimental): Topical, single application of APZ2; 500000 cells per square cm;
  Interventions: Biological: APZ2 application

INTERVENTIONS:
Biological: APZ2 application — Application of IMP on patients wound.

SUMMARY:
The aim of this clinical trial is to investigate the efficacy (by monitoring the wound size reduction) and safety (by monitoring occurring adverse events) of the investigational medicinal product APZ2 after one single application on chronic venous leg ulcer wounds.

DETAILED DESCRIPTION:
This is an interventional, single arm, phase I/IIa clinical trial to investigate the efficacy and safety of ABCB5+ mesenchymal stem cells (MSCs) on wound healing in patients with chronic venous ulcer (CVU). Autologous MSCs will be isolated ex vivo from a small skin biopsy and will be expanded in vitro. The IMP APZ2 containing the ABCB5+ cells will then be applied on the wound surface of CVU under local anesthesia.

Patients are followed up for efficacy for 3 months which allows to distinguish actual wound healing from transient wound coverage.

The wound healing process will be documented by standardized photography. The wound size evaluation will start on the day of the first change of wound dressing. The quality of the wound healing process will be assessed on the basis of formation of granulation tissue, epithelialization and wound exudation.

Pain will be assessed using a numerical rating scale and quality of life will be investigated with standardized and validated questionnaires. To assess long-term safety of APZ2 an additional follow-up visit at Month 12 post IMP application is included.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 85 years;
2. Chronic venous leg ulcer (as defined by the current AWMF guidelines: therapy resistant ulcer that shows no improvement within 3 months despite of optimal phlebological therapies or is not healed within 12 months) for at least 6 weeks but shorter than 3 years diagnosed by doppler ultrasonography (DUS), ankle brachial index (ABI, 0.9-1.3), physical examination and dermatological review;
3. Wound size between 5 and 50 square cm measured by a standardized photography at the screening visit;
4. Wound location between knee and ankle;
5. Patients suffering from 2 ulcers at the same extremity, as long as these ulcers are separated by a minimum bridge of 1 cm of epithelialized skin;
6. Patients must agree to have at least one biopsy performed before treatment. In case IMP production from the first biopsy is not successful, a second biopsy will be taken;
7. Body mass index (BMI) between 20 and 40 kg/m²;
8. Patients understand the nature of the procedure and are providing written informed consent prior to any clinical trial procedure;
9. Women of childbearing potential must have a negative blood pregnancy test at Screening and at Visit 5 before the IMP application;
10. Women of childbearing potential and their partner must be willing to use highly effective contraceptive methods during the course of the clinical trial.

Exclusion Criteria:

General exclusion criteria

1. Evidence of the ulcer extending to the underlying muscle, tendon, or bone;
2. Current long-term use (more than 14 days) of steroid medication above Cushing-threshold dose (>7.5 mg/d prednisone or equivalent);
3. Diabetes mellitus that has to be evaluated by blood test (Hemoglobin A1c [HbA1c] > 7.5%);
4. Peripheral Artery Disease (PAD) including claudication with need of treatment;
5. Acute deep vein thrombosis (maximum 30 days from diagnosis) or a still untreated deep vein thrombosis;
6. Unable to tolerate leg ulcer compression bandage;
7. Infection of the target ulcer requiring treatment as judged clinically;
8. Wound size <1.5 cm² measured by a standardized photography at Visit 5;
9. Any chronic dermatological disorders diagnosed at the investigator's discretion;
10. Skin disorders, unrelated to the ulcer, that are present adjacent to the target wound;
11. Current use of medications that influence wound healing: systemic immunosuppressives, cytotoxic medicinal products, and systemic steroids (above Cushing-threshold level);
12. Known abuse of alcohol, drugs, or medicinal products;
13. Cancerous or pre-cancerous lesions adjacent to the target wound;
14. Patients anticipated to be unwilling or unable to comply with the requirements of the protocol;
15. Pregnant or lactating women;
16. Systemic infectious disease diagnosed by serology testing for syphilis (acute), human immunodeficiency virus (HIV˗1, HIV-2), hepatitis B (acute) or C infection at Screening or at Visit 2;
17. Any known allergies to components of the IMP;
18. Prior surgical procedures such as bypass or mesh-graft treatment within 2 months prior to IMP application;
19. Treatment with active wound care agents (e.g. Iruxol, local antibiotics or silver dressings), which have not been paused 14 days before IMP application;
20. Current or previous (within 30 days of enrollment) treatment with another IMP, or participation and/or under follow-up in another clinical trial;
21. Previous participation in this clinical trial;
22. Evidence of any other medical conditions (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment;
23. Employees of the sponsor, or employees or relatives of the investigator.

Exclusion criteria for efficacy assessments

1. A wound size enlargement of more than 25% between the wound assessment at the screening visit and the wound assessment at Visit 5;
2. A wound size reduction of more than 50% between the wound assessment at the screening visit and wound assessment at Visit 5.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Percentage of wound size reduction | Week 12 post baseline, or last available post-baseline measurement if the Week 12 measurement is missing
  Percentage of wound size reduction at Week 12, or last available post-baseline measurement if the Week 12 measurement is missing (last observation carried forward [LOCF])
Assessment of adverse event (AE) occurrence | At biopsy removal, 1-3 days post biopsy, 7-10 days post biopsy, 6-12 weeks post biopsy; at baseline and days 3, 8 and weeks 2, 3, 4, 6, 8, 10, 12 and month 12 post baseline
  All during the clinical trial occurring AEs will be registered, documented and evaluated.

SECONDARY OUTCOMES:
Percentage of wound size reduction | Weeks 2, 3, 4, 6, 8, 10 and 12 post baseline
  Percentage of wound size reduction at Weeks 2, 3, 4, 6, 8, 10 and 12 (without LOCF)
Absolute wound size reduction | Weeks 2, 3, 4, 6, 8, 10, and 12 post baseline
Proportion of patients achieving complete wound closure | Weeks 2, 3, 4, 6, 8, 10, and 12 post baseline and at any time point up to week 12
Time to first complete wound closure | Between baseline and week 12 post baseline
  A priori specification not possible
Proportion of patients achieving 30% wound closure | Weeks 2, 3, 4, 6, 8, 10, 12 post baseline and at any time point up to week 12
Time to first 30% wound closure | Between baseline and week 12 post baseline
  A priori specification not possible
Percentage of wound epithelialization | At baseline and days 3, 8 and weeks 2, 3, 4, 6, 8, 10, 12 post baseline
  Amount of wound epithelialization in % of wound area will be assessed by the investigator based on image analysis of images taken from the wound.
Formation of granulation tissue and wound exudation | At baseline and days 3, 8 and weeks 2, 3, 4, 6, 8, 10, 12 post baseline
  Formation of granulation tissue in % of wound area will be assessed by the investigator based on image analysis of images taken from the wound.
  Wound exudation will be classified by the investigator using following scores:
  * High: Small amounts of fluid or free fluids are visible when the dressing is removed; dressing is extensively marked or wet
  * Moderate: Small amounts of fluid are visible when dressing is removed; wound bed may appear glossy; Primary dressing may be lightly marked
  * Low: Wound bed is dry; there is no visible moisture; Primary dressing is unmarked; dressing may be adherent to wound
Pain assessment as per numerical rating scale (NRS) | At baseline and days 1-3, 8 and weeks 2, 3, 4, 6, 8, 10, 12 post baseline
Quality of life (QoL) assessment using the SF-36 questionnaire | At baseline and weeks 4, 8, 12 post baseline
Dermatologic quality of life assessment using the DLQI questionnaire | At baseline and weeks 4, 8, 12 post baseline
Physical examination and vital parameters | At Screening, baseline, week 12, month 12

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kerstan, PD Dr.med., Principal Investigator — Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie Universitätsklinikum Würzburg
Locations (2):
- Germany (2):
  - Venenzentrum der Dermatologischen und Gefäßchirurgischen Kliniken, Kliniken der Ruhr-Universität Bochum im St. Maria-Hilf-Krankenhaus, Bochum
  - Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided